CLINICAL TRIAL: NCT01123733
Title: Breastfeeding Practice in Taiwan - Evaluation the Non-Baby-Friendly Hospitals Intervention Strategies to Breastfeeding Practice
Brief Title: Breastfeeding Practice Evaluation in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: National Taipei College of Nursing (Other)
Responsible Party: Chun-Sen Hsu, Department of obstetrics & gynecology, Taipei Medical University WanFang Hospital
Other Study IDs: 98068
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Postpartum Women
Keywords: Baby-friendly hospitals; Non baby-friendly hospitals; Breastfeeding; Ten steps for successful breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project aims to analyze and compare the prevalence of breastfeeding at one hour after delivery, discharge from hospital, one month, two months, four months, and six months after delivery and to examine factors associated with breastfeeding between baby-friendly hospitals and non baby-friendly ones. Employing a prospective cohort design, the study population is mothers who gave lived births in Taiwan area from August, 2009 to March, 2010. At least 11 hospitals both in non baby-friendly and baby-friendly hospitals from northern, middle, southern and east areas will be asked for permission to join this study (totally 22 hospitals). The research assistants will contact each eligible participant in the hospitals and explained the purposes and procedure of the study. Once permission was obtained, mothers will be asked to write a questionnaire and their telephone numbers as well as address for future contacts. After the individual case returned home, the collection of data was mainly via telephone interviews. However, if the individual case could not be contacted more than two times via telephone, she would be surveyed by questionnaire. The collection of data showed the state of mother milk feeding one month, two months, four months, or six months after delivery. 1, 000 effective questionnaires were expected to be returned (500 ones from baby friendly hospitals; 500 ones, from non baby-friendly hospitals.) The survey include questions on breastfeeding experiences (one hour after delivery, discharge from hospital, one month, two months, four months, and six months), planned duration of breastfeeding, socio-demographic information, perceived baby-friendly practices at hospital, social support regarding breastfeeding, prior infant feeding method, maternal and infant health conditions, mother's working plan, receipt of formula samples and commercial message during perinatal period. The researcher hopes that based on the research results we can have a better understanding of the influencing factors of promoting mother milk feeding in non baby-friendly hospitals, and that we know how to raise the breastfeeding rate in Taiwan area, which can serve as references for the governmental policies.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women who gave lived births in Taiwan area from August, 2009 to March, 2010.
* Be able to understand the content of questionnaire

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Postpartum women who gave lived births in Taiwan
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-05 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Sen Hsu, MD, Principal Investigator — Department of obstetrics & gynecology, Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taipei, Taiwan